CLINICAL TRIAL: NCT06094517
Title: What Are Persistent Lower Back Pain Patients' Views of Sleep Health Within an Outpatient
Brief Title: What Are Persistent Lower Back Pain Patients' Views of Sleep Health Within an Outpatient Musculoskeletal Physiotherapy Setting?
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheffield Hallam University (Other)
Collaborators: Chesterfield Royal Hospital NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: PLBP paitent view sleep Phyiso
Record Dates: First submitted 2023-10-16; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Persistent Lower Back Pain; Sleep Disturbance; Lower Back Pain; Chronic Low-back Pain
Keywords: Physiotherapy; Persistent Lower Back Pain; Sleep Disturbance; Lower Back Pain; Chronic Low-back Pain
MeSH Terms: conditions — Parasomnias; Low Back Pain | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observed Group: Patients with persistent lower back pain awaiting Physiotherapy care, undergoing interviews to assess their views of sleep health within and musculoskeletal outpatient Physiotherapy setting.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — Persistent Lower Back Pain Patients on waiting list under going a usual care pathway following referral to Physiotherapy will be interviewed for views on sleep health

SUMMARY:
The goal of this qualitative is to understand the views and opinions of patients with persistent lower back pain patients who are awaiting physiotherapy treatment with regards sleep their sleep health. The main questions it aims to answer are:

* Identify whether Patients with persistent lower back pain awaiting physiotherapy consider sleep health relevant to their condition.
* Understand whether persistent lower back pain patients awaiting physiotherapy consider sleep health within the remit of Physiotherapy?
* Understand how persistent lower back pain patients may want sleep health to be assessed or managed within an outpatient musculoskeletal Physiotherapy Setting?

Participants will undertake one semi structured interview and complete two secondary outcome measures: Pittsburgh Sleep Quality Index and Pain, Enjoyment of Life and General Activity Scale. Data will be analysed via Thematic Analysis.

DETAILED DESCRIPTION:
Background:Approximately one third of western populations suffer from sleep disturbance at least once a week and with 6-10% meeting the threshold of insomnia (National Institute of Clinical Excellence, 2022). The estimated population of the United Kingdom (UK) affected by insomnia is 37% (Morphy et al., 2007). Diminished sleep is associated with increased pain perceptions, reduced pain thresholds, physical activity levels, immune function, cognition and quality of life. Moreover, a lack of sleep correlates with increased prevalence of diabetes, obesity, cardiovascular disease, depression, and mortality (Medi, Wille & Hemels, 2017).

Over 90% of patients with Persistent Lower Back Pain (PLBP) receiving physiotherapy are affected by sleep disturbance (Roseen et al., 2020).Conventional Physiotherapy rehabilitation has shown effective in improving sleep quality in patients with PLBP as measured via Pittsburgh Sleep Quality Index (PSQI). However, Eadie et al. (2013) & Roseen et al., (2020). There is a paucity of research exploring Physiotherapies role within sleep health. Equally, studies specific to Physiotherapies role are mainly reviewed from the clinician's perspective, with a scarceness of studies providing insight into the patient perspective. To date, no studies have canvassed the opinion of patients in Physiotherapy care on the profession's role in sleep health, creating a strong footing for the proposed investigation Physiotherapist place a high value on the importance of sleep health but struggle to provide inventions citing a lack of training, resource and time. The evidence based is heavily survey based and of a quantitative nature, lacking explanation of why barriers exist, warranting further qualitative investigation (Caudwell et al. 2020 and Siengsukon, Nelson & Turkowitch 2023)

It is unclear how PLBP patients with sleep disturbance want to utilize their time in Physiotherapy care and their perceptions of Physiotherapies role within the management of sleep health (Siengsukon, Nelson & Turkowitch 2023). The proposed study would be the first to be conducted in the UK, examining PLBP patients' expectations of sleep health management within outpatient MSK physiotherapy setting.

Design and Methods:Qualitative in nature, via individual semi-structured interviews, will allow the study to explore participants' feelings and beliefs (De Jonckheere & Vaughn, 2019). The study topic is novel in design and will allow the capture of rich data and themes (Lincoln & Guba, 1985), current evidence base lacks qualitative data, especially from a patient perspective(Caudwell et al. 2020).

Recruitment and Sample Size: Recruitment will occur until the point of data saturation is reached and new themes have stopped emerging. Dickerson, Klingman & Jungquist (2016) comparable study found that interviewing 29 participants on the "Common meanings of good and bad sleep" met saturation point. Given their much wider focus, it is anticipated that interviewing 8-12 participants would meet data saturation in the proposed study. This will be reviewed for adequacy concurrently with data collection (De Jonckheere & Vaughn 2019 and Malterud, Siersma & Guassora, 2016).

Data-Collection: Semi-structured interviews will be directed by the interview guide. Transcriptions will then be reviewed and corresponded to interview notes taken to ensure accuracy. Further secondary outcome measures PSQI and Pain, Enjoyment of Life and General Activity Scale, will be collected prior to interviews via Google Forms Surveys.

Data Analysis: Data analysis will be completed by the principal investigator via a Reflexive Thematic Analysis approach.

* Dataset Familiarisation
* Data Coding
* Initial Theme Generation
* Theme Development and Review
* Theme Refining
* Writing Up

Reflexive Thematic Analysis provides a structured systematic process for the recognition of themes. It recognises the background of the research and celebrates their insight into the topic, allowing for meaningful generation of themes. Although themes should occur multiple times within the data, this approach allows for the relevance and quality of the data provided to best answer the research question as opposed to prevalence alone. To ensure rigour, prior to completing the trial practice interview with Senior Physiotherapist interested in sleep health and reviewed for appropriateness. During the interview and coding processes, a reflective log will be kept by the principal researcher, appraising their performance within the data collection and considering personal bias (Campbell et al., 2021). To ensure consistency, the interviews, initial coding and theme generation will be conducted by the Principal Investigator. Appropriateness will be reviewed by the First Supervisor.

ELIGIBILITY:
Inclusion Criteria:

* On waiting list for Outpatient MSK Physiotherapy at Chesterfield Royal Hospital NHS Foundation Trust
* PLBP (present ≥ 3 months)
* Patients ≥ 18 years

Exclusion Criteria:

* Not fluent in English
* Failure to understand study
* Previous spinal surgery
* Serous spinal pathology such as fractures or metastasis
* Inflammatory Arthritis
* Referral of pain below buttock
* Acute mental health episode

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants will be identified from self-referrals and General Practitioner (GP) referrals to outpatient Musculoskeletal Physiotherapy at Chesterfield Royal Hospital NHS Foundation Trust, Meeting the Inclusion / exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-17 (Estimated)

PRIMARY OUTCOMES:
Thematic Analysis | Completed one within 2 week of recruitment to trial
  Thematic Analysis of Data from semi structured interview

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index | Completed one within 2 week of recruitment to trial
  Self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval
Pain, Enjoyment of Life and General Activity Scale (PEG Scale) | Completed one within 2 week of recruitment to trial
  Self-rated questionnaire which assesses Pain, Enjoyment of Life and General Activity via 3 separate visual analogue scales.

IPD SHARING:
Plan to Share IPD: Undecided
Requests for anonymised core data will be considered upon request by the Principle Investigator Clive Smith ( via emails clivesmith1@nhs.net).
  Personal details will not be shared other than with responsible parties from Sheffield Hallam University or Chesterfield Royal Hospital NHS Foundation Trust in the case of concern safety concerns.

REFERENCES:
- [Background] National Institute of Clinical Excellence. (2022). Insomnia. CKS. https://cks.nice.org.uk/topics/insomnia/background-information/prevalence
- [Background] Morphy H, Dunn KM, Lewis M, Boardman HF, Croft PR. Epidemiology of insomnia: a longitudinal study in a UK population. Sleep. 2007 Mar;30(3):274-80. PMID 17425223
- [Background] Medic G, Wille M, Hemels ME. Short- and long-term health consequences of sleep disruption. Nat Sci Sleep. 2017 May 19;9:151-161. doi: 10.2147/NSS.S134864. eCollection 2017. PMID 28579842
- [Background] Roseen EJ, Gerlovin H, Femia A, Cho J, Bertisch S, Redline S, Sherman KJ, Saper R. Yoga, Physical Therapy, and Back Pain Education for Sleep Quality in Low-Income Racially Diverse Adults with Chronic Low Back Pain: a Secondary Analysis of a Randomized Controlled Trial. J Gen Intern Med. 2020 Jan;35(1):167-176. doi: 10.1007/s11606-019-05329-4. Epub 2019 Oct 30. PMID 31667747
- [Background] Eadie J, van de Water AT, Lonsdale C, Tully MA, van Mechelen W, Boreham CA, Daly L, McDonough SM, Hurley DA. Physiotherapy for sleep disturbance in people with chronic low back pain: results of a feasibility randomized controlled trial. Arch Phys Med Rehabil. 2013 Nov;94(11):2083-92. doi: 10.1016/j.apmr.2013.04.017. Epub 2013 May 2. PMID 23643716
- [Background] Lincoln, Y. S., & Guba, E. G. (1985). Naturalistic inquiry. Sage
- [Background] Caudwell, L., Himani, H., Khaw, A., Taylor, R., White, J., Rhodes, S., & Skinner, M. (2020). Attitudes and perceptions of health professionals towards sleep health: A systematic review. Physical Therapy Reviews, 25(5-6), 361-380.
- [Background] Siengsukon CF, Nelson E, Turkowitch D. Barriers and Facilitators to Implementing Sleep Health into Outpatient Physical Therapist Practice: A Survey Study. J Allied Health. 2023 Summer;52(2):e55-e61. PMID 37269038
- [Background] DeJonckheere M, Vaughn LM. Semistructured interviewing in primary care research: a balance of relationship and rigour. Fam Med Community Health. 2019 Mar 8;7(2):e000057. doi: 10.1136/fmch-2018-000057. eCollection 2019. PMID 32148704
- [Background] Dickerson SS, Klingman KJ, Jungquist CR. Common meanings of good and bad sleep in a healthy population sample. Sleep Health. 2016 Sep;2(3):253-259. doi: 10.1016/j.sleh.2016.06.004. Epub 2016 Jul 30. PMID 29073430
- [Background] Malterud K, Siersma VD, Guassora AD. Sample Size in Qualitative Interview Studies: Guided by Information Power. Qual Health Res. 2016 Nov;26(13):1753-1760. doi: 10.1177/1049732315617444. Epub 2016 Jul 10. PMID 26613970
- [Background] Campbell, K. A., Orr, E., Durepos, P., Nguyen, L., Li, L., Whitmore, C., ... & Jack, S. M. (2021). Reflexive thematic analysis for applied qualitative health research. The Qualitative Report, 26(6), 2011-2028.